CLINICAL TRIAL: NCT05925816
Title: Understanding Decision Making Using a Text-based Game
Brief Title: Guided Feedback in an Online Game Impacts Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bard College (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Justin Dainer-Best, Assistant Professor of Psychology, Bard College
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: 2021NOV10-DAI
Record Dates: First submitted 2023-06-14; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Depressive Symptoms
Keywords: depressive symptoms
MeSH Terms: conditions — Depression | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Brief interventions are conducted online and thus largely masked. All assessment is also conducted through an online survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Video (Experimental): Short video with BA intervention ideas
  Interventions: Behavioral: Video
- Active game (Experimental): Feedback Twine game
  Interventions: Behavioral: Active game
- Neutral game (Sham Comparator): Neutral Twine game
  Interventions: Behavioral: Neutral game
- No intervention (No Intervention)
- Video + Active game (Experimental): Combines Video and Active game
  Interventions: Behavioral: Video; Behavioral: Active game
- Video + Neutral game (Active Comparator): Combines Video and Neutral game
  Interventions: Behavioral: Video; Behavioral: Neutral game

INTERVENTIONS:
Behavioral: Video — Video uses BA techniques for approximately 5 minutes
  Arms: Video; Video + Active game; Video + Neutral game
Behavioral: Active game — Game provides positive feedback in response to decisions made by participants
  Arms: Active game; Video + Active game
Behavioral: Neutral game — Game without feedback
  Arms: Neutral game; Video + Neutral game

SUMMARY:
The purpose of the study is to evaluate the use of a text-based game as a way to understand decision making and knowledge related to anxiety, stress, and mood states like depression or loneliness. The investigators are interested in identifying whether participants who are given feedback before and during the game will report changes in behavior or depressive symptoms over the course of a one-week period. This is a follow-up to the published study from the researchers.

ELIGIBILITY:
Inclusion Criteria:

* 18+ age
* Eligible to participate in online research
* Able to read and respond in English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
patient health questionnaire (PHQ; 8 items) | baseline (T0) - before intervention
  The PHQ measures depression; scores range from 0 to 24 with higher scores indicating more depression.
patient health questionnaire (PHQ; 8 items) | one week following intervention (T1)
  The PHQ measures depression; scores range from 0 to 24 with higher scores indicating more depression.
Behavior in study-specific game | Completed at baseline (T0)
  For participants completing the game (neutral or active), behavior and choices made will be used as data for analyses. Game choices allow participants to decide what next activities they will "do" in the game. Analyses incorporate decision probabilities (which of 2-5 choices are selected) and compare them between conditions. The game is completed at baseline following assessment (and following video) for those assigned this arm only.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7 (GAD-7) | Baseline (T0) before intervention
  7-item measure of generalized anxiety; scores range from 0 to 21 with higher scores indicating more anxiety.
Generalized Anxiety Disorder 7 (GAD-7) | one-week follow-up (T1)
  7-item measure of generalized anxiety; scores range from 0 to 21 with higher scores indicating more anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Bard College, Annandale-on-Hudson, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and code for analyses have been shared on the Open Science Framework, https://osf.io/
Supporting Information: Study Protocol, Analytic Code
Time Frame: IPD will be available when the study is submitted for publication, beginning in 2023.
Access Criteria: Anyone will be able to access de-identified data and code.
URL: https://doi.org/10.17605/osf.io/mds4f